CLINICAL TRIAL: NCT03933163
Title: A Randomised Placebo-controlled Crossover Trial of Micronised Resveratrol as a Treatment for Friedreich Ataxia
Brief Title: Micronised Resveratrol as a Treatment for Friedreich Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36007
Record Dates: First submitted 2019-04-16; First posted 2019-05-01 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Friedreich Ataxia
Keywords: Resveratrol; Frataxin
MeSH Terms: conditions — Friedreich Ataxia | interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, placebo-controlled 2-period crossover trial of 2g/day of micronised resveratrol versus placebo. Participants will be randomised in terms of the order in which they received micronised resveratrol and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomised between receiving resveratrol in period 1 and placebo in period 2, or placebo in period 1 and resveratrol in period 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Resveratrol followed by placebo (Other): 1g micronised resveratrol twice daily for 24 weeks, a wash-out period of 4 weeks, followed by twice daily placebo for 24 weeks.
  Interventions: Drug: Resveratrol
- Placebo followed by Resveratrol (Other): Twice daily placebo for 24 weeks, a wash-out period of 4 weeks, followed by 1g micronised resveratrol twice daily for 24 weeks
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — Drug name: Micronised resveratrol. Dosage form: 500mg capsules. Alternate name: 1,3-Benzenediol, 5-[2-(4-hydroxyphenyl)ethenyl]-, (E). Ingredients: 99.50% pure trans-resveratrol. Placebo capsules will be identical in terms of taste, smell, and appearance.

SUMMARY:
The aim of this study is to assess the efficacy of micronised resveratrol as a treatment for FRDA, in terms of reducing the severity of ataxia symptoms at 24 weeks, through a randomised blinded, placebo controlled crossover trial.

DETAILED DESCRIPTION:
Friedreich ataxia (FRDA) is the most common hereditary ataxia, with an estimated prevalence in Caucasians of 1 in 30,000. Neurological features of FRDA are progressive gait and limb ataxia, absent lower limb reflexes, and loss of position and vibration sense. There are currently no treatments proven to alter the natural history of FRDA. Resveratrol is a naturally occurring compound found in red wine, berries, and nuts. It is postulated to have wide-ranging health benefits, including antioxidant, anticarcinogenic, antidiabetic and neuroprotective properties.

The study will be a double-blinded, placebo-controlled randomised 2-period crossover trial of 2g/day of micronised resveratrol in FRDA over 24 weeks. The study will enrol 40 patients with FRDA from 3 sites. The primary outcome measure is the change in modified Friedreich Ataxia Rating Scale (mFARS) score from baseline to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16 years.
2. Diagnosis of FRDA, genetically documented to be due to homozygosity for a GAA repeat expansion in intron 1 of FXN.
3. Functional stage on the Ataxia subscale of the full FARS of 1 or higher (a score of 1 is assigned if the subject has "Minimal signs detected by the physician during screening. Can run or jump without loss of balance. No disability."), and total mFARS score of ≤ 65.
4. Adequate end organ function defined as follows: (i) total bilirubin <2x upper limit of normal unless attributable to Gilbert disease, (ii) ALT and AST <1.5x upper limit of normal, (iii) Creatinine <2x upper limit of normal, (iv) neutrophils >1.5x10^9/L, (v) platelets >10^6/μL.
5. Written informed consent provided.

Exclusion Criteria:

1. Non-elective hospitalisation within the past 60 days that could be of concern in the investigator's judgment. Any hospitalisation in the previous 60 days will be assessed and if in the investigator's judgement it could compromise the individual or the study, that person will not be recruited. Examples include if the individual is hospitalised for management of cardiac morbidity such as uncontrolled arrhythmia or angina or for orthopaedic surgery for a lower limb fracture.
2. Women who are pregnant or lactating or men and women of childbearing potential who are unwilling to use contraception for the duration of the study.
3. FRDA due to compound heterozygosity for an expanded GAA repeat and a point mutation/ deletion in the FXN gene.
4. Current or recent (in last 12 months) arrhythmias including: atrial fibrillation, atrial flutter, sinus tachycardia >120/min, sinus bradycardia <50/min. Symptomatic paroxysmal arrhythmia which is recurring frequently. Cardiac insufficiency (by New York Heart Association >2). Reduced LV ejection fraction (<50%) in the last six months.
5. Medical illness that in the judgment of the investigator would jeopardise the safe completion of the study. Examples include cancer, chronic inflammatory disease, severe diabetes (type I or II, HbA1c >8%), chronic liver insufficiency, epilepsy, thrombocytosis.
6. Evidence of end organ dysfunction through failure to meet one or more parameters in inclusion criterion number 4.
7. Prior invasive cancer (excluding localised basal cell or squamous cell skin cancer).
8. Known hypersensitivity to resveratrol.
9. Use of any investigational agent within 30 days of enrolment.
10. Use of antioxidants such as vitamin E, coenzyme Q10 or idebenone within 30 days prior to enrolment.
11. Concomitant use of medications with potential for clinically relevant drug interactions. This includes medications with a narrow therapeutic range that are metabolised by the cytochrome P450 3A4, 2D6 or 2C9 systems e.g. warfarin, amiodarone.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Modified Friedreich Ataxia Rating Scale | 24 weeks
  Change in the Modified Friedreich Ataxia Rating Scale score (score range 0-99) at 24 weeks compared with baseline. Higher scores are indicative of more severe disease.

SECONDARY OUTCOMES:
Nine-Hole Peg Test | 24 weeks
  Change in the Nine-Hole Peg Test at 24 weeks compared with baseline.
Berg Balance Scale | 24 weeks
  Change in the Berg Balance Scale (score range 0-56) at 24 weeks compared with baseline. A higher score indicates lower fall risk.
Ataxia Instrumented Measure-Spoon | 24 weeks
  Change in the Ataxia Instrumented Measure-Spoon at 24 weeks compared with baseline.
Friedreich Ataxia Impact Scale | 24 weeks
  Change in the Friedreich Ataxia Impact Scale at 24 weeks compared with baseline. The Friedreich Ataxia Impact Scale comprises 8 subscales (score range 0-100) that are scored independently. A higher score indicates greater impact of Friedreich ataxia on health and well-being.
Modified Fatigue Impact Scale | 24 weeks
  Change in the Modified Fatigue Impact Scale (score range 0-24) at 24 weeks compared with baseline. Higher scores indicate a greater impact of fatigue on an individual's activities.
Measures of speech | 24 weeks
  Change in measures of speech (reading a paragraph, produce a prolonged vowel sound for 5 seconds, count from one to 20, and produce a 1-minute monologue on a pre-specified topic) at 24 weeks compared with baseline.
Measures of hearing | 24 weeks
  Change in measures of hearing using the Listening in Spatialized Noise Test (LiSN-S) at 24 weeks compared with baseline.
Cardiac parameters measured by echocardiography | 24 weeks
  Change in left ventricular global longitudinal strain at 24 weeks compared to baseline.
Cardiac parameters measured by ECG | 24 weeks
  Change in QRS duration at lead V5 at 24 weeks compared to baseline.
Frataxin levels | 24 weeks
  Change in frataxin levels at 24 weeks compared to baseline.
mRNA levels | 24 weeks
  Change in PGC-1α mRNA levels and Nrf2 mRNA levels at 24 weeks compared to baseline.
Plasma F2-isoprostane levels | 24 weeks
  Change in plasma F2-isoprostane levels at 24 weeks compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Delatycki, PhD, MBBS, Principal Investigator — Murdoch Childrens Research Institute
Locations (4):
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - University of Queensland Centre for Clinical Research, Herston, Queensland
  - Murdoch Children's Research Institute, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for analysis of the study will be available six months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by contacting martin.delatycki@vcgs.org.au.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties and there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.